CLINICAL TRIAL: NCT00796198
Title: A Pilot Study on the Effects of Cosopt on IOP Lowering and Ocular Diastolic Perfusion Pressure in Patients Not Controlled With Xalatan Monotherapy
Brief Title: Effects of Cosopt on IOP and on Ocular Diastolic Perfusion Pressure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Rolle Teresa, MD,, University of Turin, Department of di Physiopathology Clinic-Section of Ophthalmology-Eye Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COS16102007
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Glaucoma
Keywords: Glaucoma; Intraocular pressure; Ocular diastolic perfusion pressure; Dorzolamide/timolol Fixed combination; Heidelberg Retina Flowmeter
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xalatan+Cosopt (Active Comparator): Cosopt will be added to Xalatan when Xalatan is effective but not sufficient to reach the target pressure (Add group) (n = 25)
  Interventions: Drug: Xalatan+Cosopt; Drug: Xalatan
- Xalatan (Active Comparator): when Xalatan is effective and sufficient to reach the target pressure no other medication will be added (control group) (n = 25)
  Interventions: Drug: Xalatan

INTERVENTIONS:
Drug: Xalatan+Cosopt — Xalatan ophthalmic solution one drop at 10pm + Cosopt ophthalmic solution one drop at 8am and one drop at 8 pm
  Arms: Xalatan+Cosopt
Drug: Xalatan — Xalatan ophthalmic solution one drop at 10pm

SUMMARY:
Hypothesis: Studies suggest that patients with low diastolic velocity and high resistivity index in the ophthalmic artery had more progressive visual fields, the investigators hypothesize therefore that addition of Cosopt to Latanoprost could improve ocular diastolic perfusion pressure (ODPP).

Objective: To evaluate the effects of Cosopt on ODPP in patients not adequately controlled with latanoprost alone.

DETAILED DESCRIPTION:
Fifty patients with primary open angle glaucoma (POAG) treated with Xalatan for whom the monotherapy was not sufficient to achieve the target IOP, will be included in the study. Non responders were defined when IOP was > 20 mmHg or if the IOP reduction was less than 25% from the baseline IOP. Patients will be classified as having POAG when they had a typical glaucomatous visual field and/or a typical abnormal optic nerve head, open angle at gonioscopy, IOP > 21 mmHg with no treatment and no clinically apparent secondary cause for their glaucoma (EGS guidelines).

Visual fields will be assessed by an Humphrey Field Analyzer 750 (HFA, Humphrey, Inc, CA, USA), 24-2 SITA (Swedish Interactive Threshold Algorithm) standard. A glaucomatous visual field defect was defined as: 1) three adjacent points depressed by 5 dB, with one of the points depressed by at least 10 dB; 2) two adjacent points depressed by 10 dB; or 3) a 10 dB difference across the nasal horizontal meridian in two adjacent points. None of the points could be edge points unless immediately above or below the nasal horizontal meridian. In addition, visual field testing was considered reliable only when false-negative responses were less than 30% and fixation losses were less than 20% on HFA.

The abnormal optic nerve head classification was based on the presence of an optic rim notch or of diffuse / generalized loss of optic rim tissue, vertical cup/disc diameter ratio asymmetry unexplained by side differences in optic disc size, disc haemorrhage.

In each centre, patient's recruitment will start as soon as the ethical committee will approve the protocol. Each sites will recruit 10 patients (5 + 5).

Cosopt will be added to Xalatan when Xalatan is effective but not sufficient to reach the target pressure (Add group) (n = 25), while when Xalatan is effective and sufficient to reach the target pressure no other medication will be added (control group) (n = 25).

(EGS guidelines: Target pressure is a subjective value that none is able to assess (until now!). Efficacy of a drug: when the medication can decrease IOP as described in the phase three of their clinical trial. Not sufficient: when the medication is effective but is not able to reach the target IOP.)

Each patient will be submitted to three different visits:

* Baseline visit: Systemic Pressure, IOP, VF, HRF, Visual Acuity, ophthalmic examination with corneal central thickness (CCT)
* Visit at 1 month: Systemic Pressure , IOP, Visual Acuity, ophthalmic examination
* Visit at 3 months: Systemic Pressure, IOP , HRF, Visual Acuity, ophthalmic examination (+ CCT) ODPP will be calculated by: "systemic diastolic pressure - IOP" at each session.

ELIGIBILITY:
Inclusion Criteria:

* POAG patients with a pattern deviation score (or its equivalent) ranging from 2.5 dB to 6.0 dB will be included in the study. This will ensure that patients with early/mid-stage glaucoma will be homogeneously collected; avoids advanced glaucoma in which OBF may behave as a different disease state.
* Best-corrected visual acuity will be of 0.5 or better with an ametropia <5D - Dioptric transparency, non smokers.
* Age will be between 45 and 65 years.

Exclusion Criteria:n

* Normal tension glaucoma, ocular hypertension, cardiovascular and/or metabolic diseases (known to affect blood flow, as diabetes and polycythemia)
* Visual field defects other than glaucoma; use of vasoactive and/or anti-hypertensive drugs (systemic beta-blocker), use of acetazolamide
* Hypersensibility and/or contraindications to any of the molecules studied
* Previous ocular surgery
* Pregnant or nursing women and use of one of drugs for erectile dysfunction

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-06 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effects of Cosopt on ODPP in patients not adequately controlled with latanoprost alone | baseline, at 1 and 3 months

SECONDARY OUTCOMES:
To evaluate the effects of Cosopt on IOP lowering in patients not adequately controlled with latanoprost alone. | baseline, at 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Rolle, MD, Assistent Professor, Principal Investigator — University of Turin, Department of Clinical Physiopathology, Section of Ophthalmology, Eye Clinic; Teresa Rolle, MD, Assistent Professor, Principal Investigator — University of Turin, Department of Clinical Physiopathology-Section of Ophthalmology-Eye Clinic
Locations (5):
- Italy (5):
  - University of Bari, Bari
  - University of Chieti, Chieti
  - University of Genova, Genova
  - University of Siena, Siena
  - University of Turin, Turin